CLINICAL TRIAL: NCT03048305
Title: Prospective Study for Molecular Biomarkers of Normal Nasopharyngeal Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guilin Medical University, China (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof, Sun Yat-sen University
Other Study IDs: 2016-FXY-059
Record Dates: First submitted 2017-01-19; First posted 2017-02-09 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tumor tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators collect nasopharyngeal epithelium samples from healthy individuals and analyze for biomarkers compared with tumor tissues from another clinical research project. The goal of this study is to identify molecular biomarkers for prediction of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of nasopharyngeal carcinoma but excluded by biopsy

Exclusion Criteria:

* Diagnosed as nasopharyngeal carcinoma during the follow-up period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of nasopharyngeal carcinoma but excluded by biopsy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
the positive rate of risk signature in healthy individuals | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided